CLINICAL TRIAL: NCT00816179
Title: Human Clinical Trial of Diagnostic Transgastric Endoscopic Peritoneoscopy for Staging of Pancreatic Head Mass
Brief Title: Diagnostic Endoscopic Exploration for Pancreatic Head Mass
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Helical CT scans at our institution preclude the necessity for diagnostic laparoscopy in most cases at our institution.
Sponsor: Jeffrey Hazey (Other)
Collaborators: Natural Orifice Surgery Consortium for Assessment and Research (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Hazey, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007C0086
Record Dates: First submitted 2008-12-30; First posted 2008-12-31 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Pancreatic Head Mass
Keywords: Pancreatic head mass; Pancreatic cancer; NOTES; Endoscopic peritoneoscopy; Whipple; palliative gastrojejunostomy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Transgastric diagnostic endoscopic peritoneoscopy — Endoscopic abdominal exploration utilizing an endoscopically created gastrotomy.

SUMMARY:
This study is being done to find out if an endoscope passed down the throat, through the stomach, and into the abdomen can quickly and accurately examine the organs and tissue of the abdomen and take biopsies if needed.

DETAILED DESCRIPTION:
This study is being done to find out if an endoscope (a small, flexible tube with a camera mounted on the end) passed down the throat, through the stomach, and into the abdomen can quickly and accurately examine the organs and tissue of the abdomen and take biopsies if needed. We wish to determine if this endoscopic route is as fast and efficient as the laparoscopic route, which is the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-80
* Radiographic diagnosis of resectable pancreatic head mass presumed to be pancreatic adenocarcinoma

Exclusion Criteria:

* Inability to obtain informed consent
* Pregnancy
* Intra-abdominal adhesions that preclude endoscopy
* Contraindication to upper endoscopy such as stricture, stenosis of the foregut
* Previous gastric surgery
* Diagnosis of pancreatic body or tail tumor
* History or current diagnosis of gastric ulcer
* Metastatic disease diagnosed by CT, EUS, MRI, or nuclear imaging
* Patient is not a candidate for resection based upon CT, EUS, MRI, or nuclear imaging
* Antiplatelet medication not stopped at least 7 days prior to procedure
* Anticoagulant medication not stopped at least 5 days prior to procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Endoscopically visualize the abdominal cavity to determine absence or presence of metastatic lesions to successfully stage pancreatic head malignancies and direct surgical treatment. | Intraoperatively

SECONDARY OUTCOMES:
Comparison of laparoscopic exploration (retrospectively) to endoscopic exploration. | 1 year
Ability to obtain peritoneal biopsies when appropriate during transgastric endoscopic procedures. | Intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W Hazey, MD, Principal Investigator — OSUMC
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Background] Rattner D, Kalloo A; ASGE/SAGES Working Group. ASGE/SAGES Working Group on Natural Orifice Translumenal Endoscopic Surgery. October 2005. Surg Endosc. 2006 Feb;20(2):329-33. doi: 10.1007/s00464-005-3006-0. No abstract available. PMID 16402290
- [Background] White R, Winston C, Gonen M, D'Angelica M, Jarnagin W, Fong Y, Conlon K, Brennan M, Allen P. Current utility of staging laparoscopy for pancreatic and peripancreatic neoplasms. J Am Coll Surg. 2008 Mar;206(3):445-50. doi: 10.1016/j.jamcollsurg.2007.09.021. Epub 2007 Nov 26. PMID 18308214
- [Background] Lillemoe KD, Cameron JL, Hardacre JM, Sohn TA, Sauter PK, Coleman J, Pitt HA, Yeo CJ. Is prophylactic gastrojejunostomy indicated for unresectable periampullary cancer? A prospective randomized trial. Ann Surg. 1999 Sep;230(3):322-8; discussion 328-30. doi: 10.1097/00000658-199909000-00005. PMID 10493479
- [Background] Ponsky JL. Gastroenterologists as surgeons: what they need to know. Gastrointest Endosc. 2005 Mar;61(3):454. doi: 10.1016/s0016-5107(04)02632-x. No abstract available. PMID 15758924
- [Background] Wagh MS, Merrifield BF, Thompson CC. Endoscopic transgastric abdominal exploration and organ resection: initial experience in a porcine model. Clin Gastroenterol Hepatol. 2005 Sep;3(9):892-6. doi: 10.1016/s1542-3565(05)00296-x. PMID 16234027
- [Background] Merrifield BF, Wagh MS, Thompson CC. Peroral transgastric organ resection: a feasibility study in pigs. Gastrointest Endosc. 2006 Apr;63(4):693-7. doi: 10.1016/j.gie.2005.11.043. PMID 16564875
- [Background] Kalloo AN, Singh VK, Jagannath SB, Niiyama H, Hill SL, Vaughn CA, Magee CA, Kantsevoy SV. Flexible transgastric peritoneoscopy: a novel approach to diagnostic and therapeutic interventions in the peritoneal cavity. Gastrointest Endosc. 2004 Jul;60(1):114-7. doi: 10.1016/s0016-5107(04)01309-4. PMID 15229442
- [Background] Ikeda K, Fritscher-Ravens A, Mosse CA, Mills T, Tajiri H, Swain CP. Endoscopic full-thickness resection with sutured closure in a porcine model. Gastrointest Endosc. 2005 Jul;62(1):122-9. doi: 10.1016/s0016-5107(05)00517-1. PMID 15990831
- [Background] Onders RP, McGee MF, Marks J, Chak A, Rosen MJ, Ignagni A, Faulx A, Schomisch S, Ponsky J. Natural orifice transluminal endoscopic surgery (NOTES) as a diagnostic tool in the intensive care unit. Surg Endosc. 2007 Apr;21(4):681-3. doi: 10.1007/s00464-007-9214-z. Epub 2007 Feb 16. PMID 17364154
- [Background] Lima E, Rolanda C, Pego JM, Henriques-Coelho T, Silva D, Carvalho JL, Correia-Pinto J. Transvesical endoscopic peritoneoscopy: a novel 5 mm port for intra-abdominal scarless surgery. J Urol. 2006 Aug;176(2):802-5. doi: 10.1016/j.juro.2006.03.075. PMID 16813951
- [Background] McGee MF, Rosen MJ, Marks J, Chak A, Onders R, Faulx A, Ignagni A, Schomisch S, Ponsky J. A reliable method for monitoring intraabdominal pressure during natural orifice translumenal endoscopic surgery. Surg Endosc. 2007 Apr;21(4):672-6. doi: 10.1007/s00464-006-9124-5. Epub 2007 Feb 7. PMID 17285385
- [Background] Kantsevoy SV, Hu B, Jagannath SB, Vaughn CA, Beitler DM, Chung SS, Cotton PB, Gostout CJ, Hawes RH, Pasricha PJ, Magee CA, Pipitone LJ, Talamini MA, Kalloo AN. Transgastric endoscopic splenectomy: is it possible? Surg Endosc. 2006 Mar;20(3):522-5. doi: 10.1007/s00464-005-0263-x. Epub 2006 Jan 21. PMID 16432652
- [Background] Kantsevoy SV, Jagannath SB, Niiyama H, Chung SS, Cotton PB, Gostout CJ, Hawes RH, Pasricha PJ, Magee CA, Vaughn CA, Barlow D, Shimonaka H, Kalloo AN. Endoscopic gastrojejunostomy with survival in a porcine model. Gastrointest Endosc. 2005 Aug;62(2):287-92. doi: 10.1016/s0016-5107(05)01565-8. PMID 16046997
- [Background] Bergstrom M, Ikeda K, Swain P, Park PO. Transgastric anastomosis by using flexible endoscopy in a porcine model (with video). Gastrointest Endosc. 2006 Feb;63(2):307-12. doi: 10.1016/j.gie.2005.09.035. PMID 16427940
- [Background] Park PO, Bergstrom M, Ikeda K, Fritscher-Ravens A, Swain P. Experimental studies of transgastric gallbladder surgery: cholecystectomy and cholecystogastric anastomosis (videos). Gastrointest Endosc. 2005 Apr;61(4):601-6. doi: 10.1016/s0016-5107(04)02774-9. PMID 15812420
- [Background] Pai RD, Fong DG, Bundga ME, Odze RD, Rattner DW, Thompson CC. Transcolonic endoscopic cholecystectomy: a NOTES survival study in a porcine model (with video). Gastrointest Endosc. 2006 Sep;64(3):428-34. doi: 10.1016/j.gie.2006.06.079. PMID 16923495
- [Background] Jagannath SB, Kantsevoy SV, Vaughn CA, Chung SS, Cotton PB, Gostout CJ, Hawes RH, Pasricha PJ, Scorpio DG, Magee CA, Pipitone LJ, Kalloo AN. Peroral transgastric endoscopic ligation of fallopian tubes with long-term survival in a porcine model. Gastrointest Endosc. 2005 Mar;61(3):449-53. doi: 10.1016/s0016-5107(04)02828-7. PMID 15758923
- [Background] Wagh MS, Merrifield BF, Thompson CC. Survival studies after endoscopic transgastric oophorectomy and tubectomy in a porcine model. Gastrointest Endosc. 2006 Mar;63(3):473-8. doi: 10.1016/j.gie.2005.06.045. PMID 16500399
- [Background] Sclabas GM, Swain P, Swanstrom LL. Endoluminal methods for gastrotomy closure in natural orifice transenteric surgery (NOTES). Surg Innov. 2006 Mar;13(1):23-30. doi: 10.1177/155335060601300105. PMID 16708152
- [Background] Ko CW, Kalloo AN. Per-oral transgastric abdominal surgery. Chin J Dig Dis. 2006;7(2):67-70. doi: 10.1111/j.1443-9573.2006.00256.x. PMID 16643332
- See also: Home page for OSUMC Center for Minimally Invasive Surgery — http://cmis.osu.edu/